CLINICAL TRIAL: NCT04370756
Title: Beetroot Supplementation in Women Enjoying Exercise Together
Acronym: BEE SWEET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: IU Health University Hospital (Unknown); Indiana CTSI Clinical Research Center (Unknown); Bloomington Crossfit (Unknown)
Responsible Party: Principal Investigator, Stephen J. Carter, Ph.D., Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1907026303
Record Dates: First submitted 2020-04-18; First posted 2020-05-01 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Aging; Postmenopause; Obesity
Keywords: Beetroot juice; Postmenopause; Exercise training; Endothelial function
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in small (n = 4) cohorts or "waves" to facilitate social support and adherence to the supervised exercise training sessions. We anticipate having 9 waves to successfully reach our target n. This assumes that each wave will have 4 participants, hence, 4 participants x 9 waves = 36 total participants. Subsequently, participants will be randomly selected to: 1) control (EX only) or 2) EX + Beetroot Juice.
Who Masked: Participant
Masking Description: Group allocation will be determined at random using a computer-based number in blocks of 2 to ensure equal between-group distribution (i.e. n = 2 Ex only; n = 2 BR+EX). Each number will be kept in a sealed envelope until completion of Visits 1-2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ex only (Active Comparator): Participants will perform 8 weeks of supervised exercise training (EX).
  Interventions: Other: Exercise Training
- EX + BR (Experimental): Participants will perform 8 weeks of supervised exercise training (EX) plus pre-exercise consumption of beetroot juice (BR).
  Interventions: Dietary Supplement: Beetroot Juice; Other: Exercise Training

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — Participants randomly assigned to the EX + BR group will consume 140 mL beetroot juice containing approximately 12 mmol of nitrate 3 hours prior to the supervised exercise training component.
  Arms: EX + BR
Other: Exercise Training — Participants will perform 8 weeks of supervised exercise training at a frequency of 3x per week.

SUMMARY:
This study seeks to determine the feasibility of an exercise training progression with the consumption of beetroot juice prior to exercise in postmenopausal women. Results from this investigation will be used to determine preliminary effect sizes for exercise training only (control) and exercise training + beetroot juice (EX+BR) to inform the direction of larger randomized clinical trials on pre-post changes in measures of cardiovascular health and endothelial function.

DETAILED DESCRIPTION:
An increasing body of evidence has supported acute benefits of beetroot juice including lowered blood pressure and greater muscle oxygenation during exercise. Thus, consumption of beetroot juice prior to exercise may alter the perceptual difficulty for a given exercise bout -- possibly resulting in an individual exercising at a greater intensity (without the commensurate increase in discomfort). The investigators propose that repeated exposure to a relatively greater exercise stimulus (via beetroot juice) may elicit more robust cardio-metabolic adaptations compared to exercise training alone (i.e., without beetroot juice). Possible findings could inform a larger randomized clinical trial to determine if pre-exercise beetroot juice supplementation is an effective strategy to promote health related benefits.

The investigators will examine the effects of pre-exercise beetroot juice coupled with 8 weeks of supervised exercise training among post-menopausal (75 and younger) women. Qualified individuals will be required to complete an initial screening visit as well as three baseline visits (Visits 1-2). Participants will undergo a series of tests including: dual-energy X-ray absorptiometry scan, bioelectrical impedance analysis, exhaled fraction of nitric oxide, health-related questionnaires, and pulse wave velocity. Participants will also be asked to perform leg muscle function and walking tests. Following the completion of Visits 1-2, participants will attend supervised exercise training sessions 3x/week for 8 weeks. Within 2-6 days from the last exercise training session, participants will repeat the same measurement procedures.

The primary objective involves elements of feasibility (e.g., recruitment, retention, adherence, and adverse event) and to generate preliminary effect sizes for 8 weeks of exercise training for two groups: control and EX+BR. Secondary objectives involve preliminary effect sizes for pre-post changes in distance covered during the 6-minute walk test, changes in endothelial-dependent vasodilation, and biomarkers of cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women (self-report)
* Between the ages of 18-75 years (confirmed by birth date listed on participant's driver license at screening visit)
* Physician's clearance for study participation (required prior to baseline testing)
* English-speaking
* Body mass index between 25.0 to 39.9 kg/m^2 (measured on-site at screening visit)
* Able to ambulate without assistance

Exclusion Criteria:

* Unable to provide informed consent
* 18-75 of age (confirmed by birth date listed on participant's driver license at screening visit)
* Body mass index < 25.0 or >39.9 kg/m^2 (measured on-site at screening visit)
* Greater than stage II hypertension (i.e. >159/99 mm Hg)
* Current smoker (self-report)
* Currently pregnant, lactating, or trying to become pregnant (self-report)
* Habitually exercise training >= 3 times per week (self-report)
* Significant orthopedic limitations or other contraindications to strenuous exercise
* Live or work >50 miles from Bloomington study site or do not have transportation to the study site
* Anticipate elective surgery during the study period
* Plan to move residence or travel out of the local area during the study period
* History of major metabolic disease (e.g. Type I diabetes, Type II diabetes, thyroid disorders)
* Current use of anti-coagulants (e.g. Coumadin or Warfarin)
* Current use of prescription medications that affect heart rate or blood vessel dilation (e.g. phosphodiesterase-5 inhibitors, proton pump inhibitors, systemic adrenergic blockers, nitrates, calcium channel blockers, hormone replacement therapy) (self-report and confirmed on-site at screening visit)
* Psychological or social characteristic that would interfere with their ability to fully participate in the study (i.e. taking longer than allowed time to complete cognitive assessments)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 24 months
  The number of eligible participants randomized per months of recruitment time.
Retention rate | 8 weeks
  The number of randomized participants who complete at least 17 (out of 24 possible) exercise training sessions.
Adherence to exercise training intervention | 8 weeks
  The percent of exercise sessions attended out of the 24 possible sessions.
Adherence to dietary nitrate intervention | 8 weeks
  Breath analysis of fractional exhaled nitric oxide concentrations.
Perceived difficulty of training sessions | 8 weeks
  Participants will report the perceived exertion at the end of exercise sessions using the Borg category ratio-10 scale that ranges from 0 "no exertion" to 10 "maximal exertion".

SECONDARY OUTCOMES:
Distance covered during a six-minute walk test | Baseline, post-intervention
  Participants will be asked to walk as far as possible at a preferred speed for six minutes according to ATS standards. Distance covered will be measured in meters.
Soluble endothelial microparticles | Baseline, post-intervention
  Blood samples will be analyzed for adhesion molecules (sICAM-1, sVCAM-1, sE-selectin).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Carter, Ph.D., Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No IDP sharing plan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04370756/Prot_SAP_001.pdf